CLINICAL TRIAL: NCT06371027
Title: Novel Silk Fibroin Nanofiber Membrane Using Minimally Invasive Surgery in Treatment of Periodontal Intrabony Defects: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Mohamed Hamdy Hamed El-Shesheny, principle investigator. mohamed hamdy, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RECO6U/22-2022
Record Dates: First submitted 2024-04-15; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Intrabony Periodontal Defect
Keywords: intrabony defects; regenerative membranes; minimally invasive techniques; CBCT

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Minimally Invasive Surgery Technique (MIST) (Active Comparator): Minimally Invasive Surgery Technique in the area that contains an intraosseous defects with Probing depth (PD) ≥5 mm
  Interventions: Procedure: Minimally Invasive Surgery Technique (MIST)
- Minimally Invasive Surgery Technique (MIST) + Collagen Membrane (Experimental): Minimally Invasive Surgery Technique + Collagen Membrane placement in the area that contains an intraosseous defects with Probing depth (PD) ≥5 mm
  Interventions: Procedure: Minimally Invasive Surgery Technique (MIST) + collagen membrane
- Minimally Invasive Surgery Technique (MIST) + Novel Silk Fibroin (SF) nanofiber membrane (Experimental): Minimally Invasive Surgery Technique (MIST) + Novel Silk Fibroin (SF) nanofiber membrane placement in the area that contains an intraosseous defects with Probing depth (PD) ≥5 mm
  Interventions: Procedure: Minimally Invasive Surgery Technique (MIST) + Novel Silk Fibroin (SF) nanofiber membrane

INTERVENTIONS:
Procedure: Minimally Invasive Surgery Technique (MIST) + Novel Silk Fibroin (SF) nanofiber membrane — Minimally Invasive Surgery Technique (MIST) + Novel Silk Fibroin (SF) nanofiber membrane placement in the area that contains an intraosseous defects with Probing depth (PD) ≥5 mm
  Arms: Minimally Invasive Surgery Technique (MIST) + Novel Silk Fibroin (SF) nanofiber membrane
Procedure: Minimally Invasive Surgery Technique (MIST) + collagen membrane — Minimally Invasive Surgery Technique (MIST) + collagen membrane placement in the area that contains an intraosseous defects with Probing depth (PD) ≥5 mm
  Arms: Minimally Invasive Surgery Technique (MIST) + Collagen Membrane
Procedure: Minimally Invasive Surgery Technique (MIST) — Minimally Invasive Surgery Technique in the area that contains an intraosseous defects with Probing depth (PD) ≥5 mm
  Arms: Minimally Invasive Surgery Technique (MIST)

SUMMARY:
Clinically and radiographically by cone beam CT evaluate the regenerative potentials of silk fibroin (SF) nanofiber membrane, using minimally invasive surgery, for the regenerative treatment of intrabony periodontal defects.

DETAILED DESCRIPTION:
Periodontitis is a bacterially induced chronic inflammation of the periodontium that extends beyond the gingiva and involves progressive and irreversible destruction of the connective tissue attachment of the teeth.The treatment involves debridement of the tooth surface and the adjacent areas employing scaling, root planing and periodontal flap surgery. While scaling and root planing are non-surgical treatment modalities and are conservative; periodontal flap surgery gains access to the underlying bone for complete debridement achieving pocket depth reduction, periodontal regeneration, and maintenance of periodontium in healthy condition feasible by routine home care methods by the patient.

Guided tissue regeneration (GTR) therapy is playing a key role in the management of intrabony defects. Current resorbable and non-resorbable membranes act as a physical barrier to avoid connective and epithelial tissue down-growth into the defect, favoring the regeneration of periodontal tissues. However, these conventional membranes possess many structural, mechanical, and bio-functional limitations and the "ideal" membrane for use in periodontal regenerative therapy has yet to be developed. Based on a graded-biomaterials approach, we have hypothesized that a biologically active and spatially designed and functionally graded nanofibrous material that mimics closely the native extracellular matrix ECM could succeed as the next generation of GTR membranes for periodontal tissue engineering. In the current study, using a minimally invasive surgical approach, we will compare a novel silk fibroin (SF) nanofiber membrane to collagen membrane as a regenerative treatment of intrabony periodontal defects.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years old. 2. Patients with periodontitis Stage III Grade C. 3. Single-rooted and multi-rooted vital teeth in either the maxilla or the mandible. 4. Probing depth (PD) ≥5 mm at the site of intraosseous defects 4 weeks following initial therapy. 5. Periodontal 2- or 3-wall intrabony defects (IBDs), measuring ≥3 mm from the alveolar crest to the defect base, estimated by radiographic evaluation (Periapical X-ray). 6. Absence of a history of periodontal surgery at the involved sites in the last 6 months. 7. History of compliance with oral hygiene instructions and periodontal recall. 8. Full mouth plaque score and bleeding on probing score ≤20% after phase I therapy.

Exclusion Criteria:

* 1. Patients with systemic illness known to affect the outcome of periodontal therapy, including diabetes, immune deficiencies, etc.24 2. Pregnant and lactating women 3. Current use of any form of tobacco.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Novel Silk Fibroin Nanofiber Membrane using minimally invasive surgery in Treatment of Periodontal Intrabony Defects | 6 months after surgery
  The primary outcome variable in this clinical study will be the change in bone fill as measured by cone beam CT

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry O6U, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided